CLINICAL TRIAL: NCT02852070
Title: Study Bronchoalveolar Lavage Fluid Driven Pathogenic Diagnosis of Lower Respiratory Tract Infections-A Prospective Multicenter Clinical Trial (BALFinder Study)
Brief Title: Study Bronchoalveolar Lavage Fluid Driven Pathogenic Diagnosis of Lower Respiratory Tract Infections
Acronym: BALFinder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Bin Cao, Clinical professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NCT02852070
Record Dates: First submitted 2016-06-21; First posted 2016-08-02 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Lower Respiratory Tract Infections
Keywords: bronchoalveolar lavage; lower respiratory tract infections
MeSH Terms: interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Active Comparator): Bronchoscopy examination with 120ml sterile saline solution for bronchoalveolar lavage
  Interventions: Procedure: bronchoalveolar lavage 120ml
- observation group (Experimental): Bronchoscopy examination with 60ml sterile saline solution for bronchoalveolar lavage
  Interventions: Procedure: bronchoalveolar lavage 60ml

INTERVENTIONS:
Procedure: bronchoalveolar lavage 120ml — 120mL sterile saline solution instilled into the distal bronchial tree in 3 times
  Arms: control group
Procedure: bronchoalveolar lavage 60ml — 60mL sterile saline solution instilled into the distal bronchial tree in 3 times
  Arms: observation group

SUMMARY:
Comparison of microbiological yield from Bronchoalveolar Lavage Fluid (BALF) for the two common-used volume bronchoalveolar lavages(60ml and 120ml)in patients with different types of lower respiratory tract infection.

Assessment of the safety of two common-used volume bronchoalveolar lavages(60ml and 120ml), including the incidence of hospital-acquired pneumonia within 14 days after bronchoscopy, and other bronchoalveolar lavage related adverse events.

DETAILED DESCRIPTION:
The morbidity and mortality of lower respiratory tract infection gradually increased in recent years, but the etiological diagnosis rate is still low. Quickly identifying the pathogenic bacteria and the corresponding antimicrobial therapy treatment is particularly important. Fibrotic bronchoscopy combined with bronchoalveolar lavage (BAL) has become a routine diagnostic tool for pulmonary infections in immunocompromised patients.

The correct operation of bronchoalveolar lavage and normalization of bronchoalveolar lavage fluid is a prerequisite for the exact results of the pathogen of BALF.

American Thoracic Society recommended amount of 100-300ml of saline solution was instilled into the distal bronchial tree in the diagnosis of interstitial lung diseases. But there is no standard of lavage fluid volume in the etiological diagnosis of lower respiratory tract infections, ranging from 60ml to 250ml ever reported in literature.

Less lavage volume would be more safer in patients with lower respiratory tract infections. The investigators hypothesize that microbiological yield would be no significant difference in patients with low volume （60ml) compared with large volume (120ml).

The purpose of this study is to explore a more effective and safer way of bronchoalveolar lavage in lower respiratory tract infection patients, and determine the pathogenic distribution among them.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of lower respiratory infection
2. Indication for bronchoalveolar lavage.

Exclusion Criteria:

1. Noninfectious pulmonary infiltration
2. Contraindication of bronchoscopy： Severe heart or pulmonary dysfunction Recent occurrence of myocardial infarction unstable angina pectoris Severe coagulation disorders (DIC), Massive hemoptysis Gastrointestinal bleeding Thrombocytopenia (<50*109/L) Severe superior vena cava obstruction syndrome Aortic aneurysm Multiple pulmonary bulla Extreme exhaustion
3. Diagnosed or highly suspected of tuberculosis infection
4. Researchers think that can not be entered into the group.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-01 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Microbiological yield | 2 years
  Comparison of microbiological yield of two arms with different BALF volume in patients with lower respiratory tract infection in a multicenter, prospective, randomized, single blind study

SECONDARY OUTCOMES:
Sensitivity and specificity of BALF galactomannan test in the diagnosis of invasive pulmonary fungal infections | 2 years
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 years
  Compare the safety of two groups included incidence of hospital acquired penumonia within 14 days after bronchoscopy, and vital signs, oxygenation, and laboratory tests before and after lavage
Sensitivity and specificity of PCR-based microbiological tests | 2 years
  Microbiological spectrum of pneumonia diagnosed by PCR, as compared with traditional microbiological methods

CONTACTS AND LOCATIONS:
Overall Officials: Cao Bin, MD, Study Chair — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No